CLINICAL TRIAL: NCT07058155
Title: OPTIMAL Trial: Optimizing Portal Hypertension With TIPS and Interval Metabolic Surgery for Advanced Liver Disease
Brief Title: Optimizing Portal Hypertension With TIPS and Interval Metabolic Surgery for Advanced Liver Disease
Acronym: OPTIMAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Ali Aminian, MD (Unknown)
Responsible Party: Principal Investigator, Sobia N. Laique, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-421
Record Dates: First submitted 2025-06-27; First posted 2025-07-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Liver Cirrhoses; Portal Hypertension Related to Cirrhosis; Severe Obesity; TIPS
Keywords: Sleeve Gastrectomy; Transjugular Intrahepatic Portosystemic Shunt (TIPS); Bariatric Surgery / Metabolic Surgery; Clinically Significant Portal Hypertension (CSPH); Health-Related Quality of Life (HRQOL); SF-36 Questionnaire; Weight Loss; Metabolic Dysfunction-Associated Steatohepatitis (MASH); Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD); Randomized Controlled Trial
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Topiramate; Phentermine; Glucagon-Like Peptide-1 Receptor Agonists; Diet Therapy

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial (1:1) comparing pre-operative TIPS followed by sleeve gastrectomy (TIPS + SG) versus best-option medical weight management in adults (BMI ≥ 35-70 kg/m²) with compensated cirrhosis and clinically significant portal hypertension.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIPS + Sleeve Gastrectomy (Experimental): Participants first undergo transjugular intrahepatic portosystemic shunt (TIPS) placement (target HVPG < 12 mmHg or ≥ 50 % reduction). After portal pressure stabilization-ideally 4-6 weeks, allowed ≤ 6 months-they receive laparoscopic or robotic sleeve gastrectomy. Standard peri- and post-operative care, plus routine lifestyle counseling, are provided.
  Interventions: Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS); Procedure: Sleeve Gastrectomy; Behavioral: Lifestyle Counseling - Diet & Physical-Activity Program
- Best-Option Medical Weight Management (Active Comparator): Participants will follow an individualized, clinician-directed medical weight loss program that includes dietary and physical activity counseling, behavior modification strategies, and best available anti-obesity pharmacotherapy (e.g., GLP-1 receptor agonists, dual incretin agonists, first generation AOMs).
  Interventions: Drug: Anti-Obesity Pharmacotherapy (Class Effect); Behavioral: Lifestyle Counseling - Diet & Physical-Activity Program

INTERVENTIONS:
Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS) — Fluoroscopically guided placement of a covered stent creating a portosystemic shunt between hepatic and portal veins. Goal: ≥ 50 % HVPG reduction or final HVPG < 12 mmHg. Conducted 4-6 weeks (≤ 6 months allowed) before bariatric surgery; standard post-TIPS surveillance ultrasound and EGD to confirm patency and variceal resolution.
  Other Names: TIPS
  Arms: TIPS + Sleeve Gastrectomy
Procedure: Sleeve Gastrectomy — Longitudinal resection of ~80 % of stomach via laparoscopic or robotic approach, preserving pylorus. Performed after successful TIPS once portal pressures stabilize (< 6 months post-TIPS). Standard peri-operative care, micronutrient supplementation, and bariatric follow-up per ASMBS guidelines.
  Other Names: SG
  Arms: TIPS + Sleeve Gastrectomy
Drug: Anti-Obesity Pharmacotherapy (Class Effect) — Clinician-selected, evidence-based anti-obesity medications (AOMs) used at the treating provider's discretion. Agents may include incretin-based therapies (e.g., Semaglutide, Tirzepatide) or other FDA-approved AOMs such as Topiramate or Phentermine. Dosing and titration follow standard labeling; no specific drug is mandated. The study assesses the overall class effect of pharmacotherapy rather than any single agent.
  Other Names: GLP-1 receptor agonist; Topiramate; Phentermine; Incretin Mimetics
  Arms: Best-Option Medical Weight Management
Behavioral: Lifestyle Counseling - Diet & Physical-Activity Program — Regular sessions with a registered dietitian or equivalent (in-person or virtual) focusing on adherence to a reduced-calorie diet, structured physical-activity regimen, and behavior-change strategies. Counseling occurs throughout the 6-month study period and is considered standard care for this patient population.
  Other Names: Dietary modification; Exercise counseling; Behavioral weight-loss coaching

SUMMARY:
Cirrhosis is a form of advanced liver disease that can lead to serious complications, especially when combined with severe obesity. Many patients with cirrhosis also develop a condition called clinically significant portal hypertension (CSPH), which is increased pressure in the veins of the liver. CSPH raises the risk of life-threatening events like internal bleeding and liver failure. Unfortunately, treatment options for people who have both cirrhosis and severe obesity are very limited, especially when portal hypertension is present.

This study, called the OPTIMAL Trial, is a randomized clinical trial designed to evaluate whether combining two procedures improves health outcomes in this high-risk population. The first procedure, called TIPS (Transjugular Intrahepatic Portosystemic Shunt), is a minimally invasive treatment that reduces pressure in the liver by creating a pathway for blood to flow more easily. The second procedure is sleeve gastrectomy, a form of metabolic (bariatric) surgery that helps patients lose weight and improve related conditions like diabetes.

The study will compare two groups:

1. One group will receive TIPS followed by sleeve gastrectomy (TIPS+SG).
2. The other group will receive medical weight management (standard non-surgical care, including diet, lifestyle changes, and weight loss medications).

All participants will have severe obesity and cirrhosis with CSPH but will not have decompensated liver disease (such as large amounts of fluid in the abdomen, a history of variceal bleeding, or recent liver failure). Eligible participants will be randomly assigned to one of the two groups.

The main goal of the study is to determine whether the combination of TIPS + SG improves quality of life and leads to greater weight loss compared to medical therapy alone. The study will also monitor for any complications from either the procedures or the medical treatment.

Participants will be followed for 6 months after their treatment starts, with periodic assessments of their physical health, liver function, and overall well-being. Some participants may also be followed for a longer period to assess long-term outcomes.

This study hopes to provide high-quality evidence for a novel, stepwise treatment strategy that may help people with obesity and liver disease live longer, healthier lives. If successful, it could change how advanced liver disease and obesity are managed together, especially in patients who currently have few safe and effective options. All study care is provided at Cleveland Clinic, Cleveland, Ohio, USA.

DETAILED DESCRIPTION:
Obesity and metabolic dysfunction-associated steatotic liver disease (MASLD) are now among the leading global causes of cirrhosis. Up to one-third of individuals with cirrhosis also have class II or III obesity, which exacerbates portal hypertension, accelerates liver disease progression, and can limit eligibility for liver transplantation. Metabolic (bariatric) surgery is an established treatment that induces sustained weight loss and improves metabolic and hepatic outcomes. However, the presence of clinically significant portal hypertension (CSPH) increases the risks of surgery, including intraoperative bleeding and postoperative hepatic decompensation. Small retrospective studies suggest that placing a transjugular intrahepatic portosystemic shunt (TIPS) before surgery may reduce these risks by decompressing the portal venous system. To date, no prospective randomized trial has evaluated this approach.

The OPTIMAL Trial (Optimizing Portal Hypertension with TIPS and Interval Metabolic Surgery for Advanced Liver Disease) is a single-center, prospective randomized controlled trial designed to determine whether a staged strategy using TIPS followed by sleeve gastrectomy improves health-related quality of life (HRQoL), weight loss, and safety in patients with cirrhosis, severe obesity, and CSPH compared to medical management alone.

The trial will enroll 70 adults aged 18 to 70 years with a body mass index (BMI) between 35 and 70 kg/m², biopsy-proven or elastography-confirmed cirrhosis, and objective evidence of CSPH. Inclusion criteria include Child-Pugh class A or B liver function, MELD 3.0 score <=15, and platelet count >= 50,000 /µL. Key exclusion criteria include decompensated cirrhosis, defined as moderate-to-large volume ascites, hepatic encephalopathy, or patients undergoing liver transplant evaluation. Patients with a history of variceal hemorrhage or small-volume ascites may still be eligible. Other exclusions include MELD 3.0 > 15, portal vein thrombosis, hepatocellular carcinoma, prior metabolic surgery, pregnancy, active substance use, untreated psychiatric illness, and severe cardiopulmonary disease that would preclude surgery or anesthesia.

After informed consent, participants will be randomized in a 1:1 ratio to one of two arms. The intervention group will undergo TIPS placement, aiming for at least a 50 percent reduction in hepatic venous pressure gradient (HVPG) or a final HVPG less than 12 mmHg, followed by sleeve gastrectomy approximately 4 to 6 weeks later. The control group will receive structured lifestyle counseling and, when clinically indicated, FDA-approved pharmacologic therapies for weight management and diabetes.

Follow-up visits at 1, 3, and 6 months will assess weight, vital signs, adverse events, and MELD 3.0 laboratory values. Liver Doppler ultrasound will be performed in the intervention group to assess TIPS patency per standard of care. Both groups will complete the SF-36 survey to evaluate health-related quality of life. The primary outcome is the change in SF-36 Physical Component Summary (PCS) score from baseline to 6 months. Secondary outcomes include percentage of total body weight loss, incidence of serious liver-related complications such as hepatic encephalopathy, variceal bleeding, and acute-on-chronic liver failure, as well as changes in SF-36 scores at 1 and 3 months. Exploratory outcomes include changes in MELD 3.0 parameters (bilirubin, albumin, INR, sodium, and creatinine); proportion of participants achieving 5% to 25% weight loss; changes in BMI, waist circumference, and body composition; changes in glucose and HbA1c in patients with type 2 diabetes; proportion meeting HbA1c targets (<6.5% without medications, <7% overall); and changes in cardiovascular and diabetes medication use.

Following randomization, all patients who receive TIPS or start nonsurgical management will be analyzed based on the intention-to-treat plan. Furthermore, patients who undergo TIPS placement but not sleeve gastrectomy for any reason, such as the development of de novo portal vein thrombosis, development of de novo acute renal failure, or persistent esophageal varices, will not be included in the per-protocol (on treatment) analysis.

This trial will generate the first prospective data evaluating whether a combined approach of portal pressure reduction and metabolic surgery can safely and effectively improve quality of life, metabolic control, and liver-related outcomes in patients with cirrhosis, severe obesity, and CSPH.

ELIGIBILITY:
Inclusion Criteria

1. Candidate for general anesthesia.
2. Age 18-70 years at consent.
3. BMI 35-70 kg/m² at first study visit.
4. Eligible for sleeve gastrectomy per ASMBS/IFSO 2022 guidelines.
5. Insurance coverage for metabolic surgery.
6. Current or prior anti-obesity medication use permitted.
7. Liver cirrhosis confirmed by biopsy or non-invasive assessment.
8. Clinically significant portal hypertension (HVPG ≥ 10 mm Hg, or esophagogastric varices / portal-hypertensive gastropathy, or imaging evidence of collaterals/dilated portal vein).
9. Able and willing to provide informed consent and comply with study procedures.
10. Women of child-bearing potential: negative urine pregnancy test at screening and randomization and agreement to reliable contraception for 2 years.

Exclusion Criteria

1. Prior bariatric/metabolic surgery (except removed devices ≥ 3 months earlier).
2. Prior complex foregut surgery.
3. History of solid-organ transplant.
4. Severe pulmonary disease (FEV1 < 50 % predicted).
5. Significant cardiac or atherosclerotic disease with planned re-vascularization within 12 months.
6. ASA class IV or V uncompensated cardiopulmonary disease.
7. Left-ventricular ejection fraction < 25 % or MI/unstable angina/stroke/heart surgery/coronary stent within 6 months.
8. Hiatal hernia > 7 cm or LA grade C/D erosive esophagitis.
9. Active Crohn's disease.
10. Severe psychiatric illness, dementia, active psychosis, history of suicide attempt, or alcohol/substance abuse within 12 months.
11. Pregnant, breastfeeding, planning pregnancy, or not using adequate contraception.
12. Malignancy within the prior 12 months (except non-melanoma skin cancer).
13. Life expectancy < 2 years in investigator's judgment.
14. Investigational therapy within 3 months.
15. Acute pancreatitis ≤ 90 days.
16. Portal vein thrombosis at screening.
17. Decompensated cirrhosis (moderate/large ascites, hepatic encephalopathy, or listed for liver transplant); small ascites or prior variceal bleed allowed.
18. Total bilirubin > 3 mg/dL, INR > 1.7, or platelets < 50 000/µL (within 1 month).
19. Significant alcohol intake (> 14 units/week women, > 21 units/week men) within the prior 12 months.
20. eGFR < 45 mL/min/1.73 m² or on dialysis (within 1 month).
21. AIDS.
22. Unable to understand study or give consent.
23. Plans to move more than 3 hours from Cleveland within 6 months.
24. Previous randomization in this trial.
25. Any condition that, in the investigator's opinion, places the subject at undue risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in SF-36 Physical Component Summary (PCS) Score From Baseline to 6 Months | At 6 months after treatment initiation (Day 0 = TIPS placement date or start of medical management).
  Difference between baseline and 6-month SF-36 PCS score (0-100 scale; higher values = better physical health-related quality of life). Positive change denotes improvement.

SECONDARY OUTCOMES:
Percent Total Body-Weight Loss (%TBWL) at 6 Months | At 6 months after treatment initiation
  %TBWL = ((baseline weight - 6-month weight) ÷ baseline weight) × 100.
Incidence of Serious Complication Composite Within 6 Months | Up to 6 months after treatment initiation
  Proportion of participants experiencing ≥ 1 of the following: severe hepatic encephalopathy (requiring hospitalization/intubation/TIPS revision), variceal hemorrhage, acute-on-chronic liver failure, deep intra-abdominal infection, severe sepsis, blood transfusion, pulmonary embolism, initiation of dialysis, or death.
Change in SF-36 Physical Component Score From Baseline to 1 Month | Baseline and 1 month
  Differences in SF-36 Physical Component Score at one month versus baseline (higher = better physical health-related quality of life).
Change in SF-36 Mental Component Score From Baseline to 1 Month. | Baseline and 1 month.
  Differences in SF-36 Mental Component Score at one month versus baseline (higher = better mental health-related quality of life).
Change in SF-36 Physical Component Score From Baseline to 3 Months | Baseline and 3 months
  Differences in SF-36 Physical Component Score at three months versus baseline (higher = better physical health-related quality of life).
Change in SF-36 Mental Component Score From Baseline to 3 Months. | Baseline and 3 months.
  Differences in SF-36 Mental Component Score at three months versus baseline (higher = better mental health-related quality of life).

OTHER OUTCOMES:
Change in HbA1c (%) | Baseline and 6 months (Week 24) after treatment initiation
  Mean absolute change in glycated hemoglobin (HbA1c, percent) between baseline and each follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Laique, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No